CLINICAL TRIAL: NCT03547141
Title: A Randomized, Double-blind, Active-controlled, Single-center, Phase 1 Study to Determine the Pharmacodynamic and Safety of MBA-P01 in Healthy Male Volunteers
Brief Title: Pharmacodynamic and Safety of MBA-P01 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MT14-KR18EDB102
Record Dates: First submitted 2018-04-29; First posted 2018-06-06 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- botulinum toxin 1U (Experimental)
  Interventions: Drug: MBA-P01; Drug: BOTOX
- botulinum toxin 5U (Experimental)
  Interventions: Drug: MBA-P01; Drug: BOTOX
- botulinum toxin 15U (Experimental)
  Interventions: Drug: MBA-P01; Drug: BOTOX
- botulinum toxin 30U (Experimental)
  Interventions: Drug: MBA-P01; Drug: BOTOX

INTERVENTIONS:
Drug: MBA-P01 — injection of MBA-P01 into the muscle of each contralateral foot in equal doses
Drug: BOTOX — injection of BOTOX into the muscle of each contralateral foot in equal doses

SUMMARY:
To determine the pharmacodynamic and safety of MBA-P01 in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged between 20 and 45 years

Exclusion Criteria:

* Subjects not appropriate for participating in this study according to the investigator's opinion

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
to estimate the pharmacodynamic aspects of muscle | day 3, 14, week 4, 8, 12
  percentage of reduction of CMAP amplitude of the muscle from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Myungeun Chung, Principal Investigator — The Catholic University, St. Paul's Hospital
Locations (1):
- The Catholic University of Korea, St. Paul's Hospital, Seoul, South Korea